CLINICAL TRIAL: NCT03464331
Title: Effectiveness of a Smartphone App in Promoting Zero-time Exercise and Fitness in Patients With Coronary Heart Disease: a Pilot Randomized Controlled Trial
Brief Title: Promoting Zero-time Exercise in Patients With Coronary Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Po-Tai Noel, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HKUCTR-2165
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Exercise Adherence

STUDY DESIGN:
Intervention Model Description: Simple individual randomization method by sequentially numbered, opaque sealed envelopes (SNOSE) will be used to ensure the research staff / interventionists and participants will be concealed from the allocation sequence. The statistician will prepare about 150 identical, opaque, sealed, A5-sized envelops, with a unique 3-digit serial number on the cover of each envelope as an identifier. Half of them will each contain a card indicating EXP and the other half, CON. For EXP, the card will further indicate activity tracker or no tracker, in 1:1 ratio. After consent, the RS will open an envelope according to the sequence of the serial number and assign participant to either EXP or CON group. The envelop must be opened according to the serial number. All others will not know the group allocation before the envelope is opened. Frequent checks (at least weekly) of these numbers will be done to ensure no deviation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXP group (Experimental): Participants in EXP group (EXP) will be asked to practise Zero-time exercises (ZTE) at least 20-30 minutes per day, and on most and preferably all days of the week.
  Interventions: Behavioral: Zero-time exercises
- CON group (Placebo Comparator): Participants in CON group (CON) will be asked to practise relaxation exercises (RE) and deep-breathing exercises (DBE) at least 30 mins every day.
  Interventions: Behavioral: relaxation exercises and deep-breathing exercises

INTERVENTIONS:
Behavioral: Zero-time exercises — The Investigators/research staff (RS) will help EXP download, operate the Zero-time exercises (ZTE) app and ZTE e-diary. The EXP can enter their goal for the chosen exercise by setting the target duration or number of completed repetitions, review their previous record, and compare their exercise frequency and time ranking with those of the other EXP. After the EXP uploads the goal and results to the ZTE e-diary, the data will be automatically sent to the ZTE app database for data analysis. The EXP will be given a paper diary to record their Zero-time exercises (ZTE). Twenty-five EXP will be given activity trackers (e.g. Fitbit) to record their steps/motion throughout the 3 months.
  Arms: EXP group
Behavioral: relaxation exercises and deep-breathing exercises — The Investigators/RS will teach the CON group (CON) to do relaxation exercises (RE) and deep-breathing exercises (DBE) for at least 30 mins every day. They will be helped download and use the electronic diary (CON_e-diary) to record their RE and DBE. The CON will also be given a paper diary to record RE and DBE they have done if they prefer to use paper diary.
  Arms: CON group

SUMMARY:
Background Physical activity (PA), is an effective means of protecting against cardiovascular disease (CVD) development. PA refers to any skeletal muscle bodily movement that requires energy expenditure. Research shows that low- to moderate-intensity muscle endurance exercise, such as walking or brisk walking for about 15-20 minutes per day, is associated with a significantly lower CVD risk regardless of body mass index. Mobile technologies such as smartphone physical exercise apps offer a potentially cost-effective platform for facilitating regular exercise, allowing individuals to set goals, receiving feedback on achievements and health information for facilitating regular exercise. "Zero-time Exercise" (ZTE) is a new concept for physical activities (PA) and exercise promotion and can easily attract attention especially when most people believe that extra time is needed to do exercise. ZTE can be done easily during most time of day, while sitting, standing, walking or waiting. These include simple movements, such as stretching and resistance (endurance) movements of the head, neck and shoulders, chest and abdominal muscles and the upper and lower limbs. When ZTE is integrated into daily life and sustained with increasing intensity, the effects could be substantial, especially for those who are sedentary and have difficulties to meet the minimal requirements of 150 minutes of at least moderate PA per week. The term is also intended to motivate people to start with simple exercises (the 'Foot-in-the-door' approach), change the mindset (that exercises need much time, money and sweats) and overcome the inertia from a sedentary lifestyle to become more active. It could also be a way to promote mental health (such as increasing happiness) through PA or exercises and enjoying the fun and satisfaction from the rapid improvements in fitness performances. Having brought some easily observable benefits quickly to those who are willing to try for a few days, ZTE might lead to more intensive or vigorous exercises requiring extra time for greater benefits.

Objective:

To test the feasibility [recruitment, dropout, and adherence to PA] of using whatsapp as an inertia reminder to promote the adherence of Zero-time Exercises (ZTE) in patients with CHD.

DETAILED DESCRIPTION:
Methods:

A 12-week single-blind randomised control design pilot study. 100 participants aged 18-69 years or above with proven stabilized acute coronary heart disease, physical inactive and having own smartphone with adequate internet technology literacy to operate the smartphone app and able to read and understand Chinese were recruited from the outpatient Cardiac Clinic in 3 hospitals.

The intervention group will be asked to practise ZTE either using the smartphone app or a zerotime exercise booklet with a focus on exercise adherence to at least 20-30 minutes per day, and on most and preferably all days of the week. The control group (CON) were asked to do deep breathing exercise at least 20 minutes daily. The exercise adherence of 25 participants in each EXP and CON groups are measured by activity trackers.

A mobile electronic whatsapp message was used as an anti- inertia reminder (AIR) to promote ZTE adherence. We used pictures with simple exercises to remind the participants in intervention group (EXP) to do ZTE regularly. Whatsapp reminders on deep breathing exercises are sent to CON. The frequency, format, whatsapp feedback and response to enquiry are the same as for EXP.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-69 years;
* Stable CHD;
* Able to walk at normal speed for at least 15 min with no breathlessness;
* Have own smartphone and can operate a smartphone app;
* Have not downloaded and used the ZTE mobile app;
* Able to read and understand Chinese;
* Willing to come back at 3-month FU (the second face-to-face session, S2) for the measurements and/or intervention

Exclusion Criteria:

* Presence of medical conditions that might limit ability to perform moderate-intensity PA;
* Currently engaging in more than 150 minutes/week of moderate/vigorous PA
* Had revascularisation performed within past 3 months;
* Currently participating in another clinical trial and/or cardiac rehabilitation programme;
* Experience wearing an activity tracker;
* Experience using a smartphone app for exercises;
* Not a Hong Kong resident, or cannot communicate in Cantonese or Putonghua.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10-18 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to the zero time exercise intervention | 3 months
  Adherence to zero time exercise intervention is calculated as the total time (duration) of ZTE done per week (as reported by participants) divided by total time (150 minutes per week as prescribed by the research team) of ZTE to be done per week. Seventy percent is considered as a good adherence rate.

CONTACTS AND LOCATIONS:
Overall Officials: Po Tai Chan, Principal Investigator — School of Nursing, HKU
Locations (3):
- China (3):
  - Grantham Hospital, Hong Kong
  - Pok Oi Hospital, Hong Kong
  - Ruttonjee Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers due to confidentiality.

REFERENCES:
- [Derived] Chan NPT, Lai AYK, Choy HK, Cheung DYT, Wan ANT, Cheng VYH, Chan KY, Lau YK, Yung CY, Cheung GOC, Lam TH. Feasibility and Potential Effectiveness of a Smartphone Zero-Time Exercise Intervention for Promoting Physical Activity and Fitness in Patients With Coronary Heart Disease: A Pilot Randomized Controlled Trial. Front Public Health. 2022 Jul 14;10:865712. doi: 10.3389/fpubh.2022.865712. eCollection 2022. PMID 35910893